CLINICAL TRIAL: NCT00125476
Title: Training and Diastolic Function in Postmenopausal Women
Brief Title: Effects of Exercise Training on Diastolic Heart Function in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 235; R21HL077165 (NIH)
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Heart Failure, Congestive; Cardiovascular Diseases
Keywords: Postmenopause
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases | interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
This study is a prospective follow-up study to the Dose-Response to Exercise in Women (DREW) study. In DREW, 450 overweight, sedentary postmenopausal women were randomly assigned to either a non-exercise control group or to 1 of 3 weekly physical activity groups. The DREW study is evaluating the dose-response of exercise training in regard to changes in multiple cardiac risk factors. This study will measure diastolic heart function in a subset of the DREW population in order to examine the relationship between dose response, changes in physical activity, and diastolic function. Diastolic heart function will be assessed using both traditional and novel echocardiographic measures.

DETAILED DESCRIPTION:
BACKGROUND:

Congestive heart failure (CHF) has become the number one reason for hospitalization in the United States. Diastolic heart dysfunction is becoming increasingly recognized as a significant factor in the etiology of CHF. Of the total affected population, 70% of patients with diastolic heart failure are female, the majority of which are elderly. There is currently no effective pharmacological therapy for the treatment of diastolic heart dysfunction. Existing cross-sectional studies and limited training trials supporting the hypothesis that exercise may improve diastolic function have only studied men. There is a need for more properly controlled and adequately powered studies examining the effect of exercise training on diastolic function, particularly in populations at high risk for CHF, such as sedentary, postmenopausal women with elevated blood pressure.

DESIGN NARRATIVE:

A total of 215 sedentary, postmenopausal women at moderate risk for cardiovascular disease will be randomly assigned to receive either exercise training or no exercise for six months. This study will measure diastolic heart function using novel echocardiographic measurements, such as pulmonary vein flow pattern, tissue Doppler, and color M-mode mitral inflow propagation velocity. The study will also measure the left ventricular mass.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive for 6 months prior to study entry; defined as sedentary and having an energy expenditure of less than 35 kcal(kgˉ¹)(dayˉ¹)
* Postmenopausal and fits one of the following criteria: over 55 years old and no natural menses for at least 5 years; less than 55 years old and no natural menses for at least 2 years and a serum follicle stimulating hormone (FSH) level greater than 40 mIU/ml; hysterectomy with documentation of bilateral oophorectomy; less than 55 years old with a hysterectomy but no documentation of bilateral oophorectomy and with an FSH level greater than 40 mIU/ml and estradiol level less than 25 pg/ml
* If taking hormone replacement therapy, must have been on a stable dose for at least 6 months, and must maintain the same dosage of the same medication throughout the study
* Body mass index between 25 and 40 kg/m²
* Systolic blood pressure between 120 and 159 mm Hg and diastolic blood pressure no greater than 99 mm Hg
* Fasting plasma glucose level less than 126 mg/dl
* Physically capable of exercise

Exclusion Criteria:

* Currently taking any antihypertensive medications
* Current or history of significant cardiovascular diseases or disorders, including arrythmias; myocarditis; cardiomyopathy; congestive heart failure; stroke or transient ischemic cerebral attacks; peripheral vascular disease with intermittent claudication; acute, chronic, or recurrent thrombophlebitis; and Stage II or III hypertension
* Current or history of total cholesterol level of at least 240 mg/dl with LDL-C level of at least 160 mg/dl or triglyceride levels of at least 300 mg/dl
* Current or history of hematologic disorders, including anemias, bleeding disorders, chronic thrombotic disorders, or hypercoagulable states
* Recent blood donation within the 6 weeks before study entry (participants also will be asked to refrain from blood donation during the study)
* Weight loss of 20 or more kilograms within the year prior to study entry
* Hospitalization for mental illness within 5 years of study entry or score of at least 10 on the Center for Epidemiological Studies Depression scale (CESD)
* Plans to be out of the city for more than 4 weeks over the next 6 months
* Other significant medical conditions, including the following: chronic or recurrent respiratory, gastrointestinal, neuromuscular, neurological, or psychiatric conditions; musculoskeletal problems interfering with exercise; autoimmune or collagen vascular diseases; immunodeficiency diseases or a positive HIV test; malignancies within 5 years of study entry, with the exception of skin cancer that is therapeutically controlled; endocrine and metabolic disorders; or any other medical condition or disease that is life-threatening or that may interfere with or be aggravated by exercise

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215
Dates: Start 2004-07

PRIMARY OUTCOMES:
Diastolic function as assessed by mitral inflow filling pattern (E/A ratio) (measured at Month 6)

SECONDARY OUTCOMES:
Pulmonary vein flow pattern
Tissue Doppler
Color M-mode mitral inflow propagation velocity
Left ventricular mass (measured at Month 6)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Blair, Study Chair — The Cooper Institute
Locations (1):
- The Cooper Institute, Dallas, Texas, United States